CLINICAL TRIAL: NCT04430270
Title: Ethical Committee at Researches of Ege University
Brief Title: Perceptions of Orthopedic Prespecialists on Patient-Specific 3D Models.
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Figen GOVSA, Prof. Dr, Senior investigator, Ege University
Other Study IDs: EGE18-5/41
Record Dates: First submitted 2020-06-03; First posted 2020-06-12 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Educational Problems
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Comparison of Perceptions of X-ray, CT and 3D Model: The study group consisted of 11 orthopaedic residents of University Hospital. Selection criteria for the 4 cases was the involved patients who required orthopaedic surgery. 4 cases for orthopaedic procedures were determined with the consensus of experts. As data collection tool was used to evaluate the perceptions of each of these imaging methods in terms of their usefulness in seeing the surgical problem, their efficiency in differential diagnosis and presurgical planning. CT images were converted into in the 3D model was prepared. The survey utilized by our group, addressed the issues in understanding bone anatomy, seeing pathology, and preparation for unexpected events. A multi-item survey was prepared to assess fellow's perception of residency training. Residents who completed their examination in the stations answered the questions on a scale of 10. Descriptive statistics and Friedman test were used for comparison analysis using IBM SPSS Statistics, version 24.
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey — Sequential Assignment

SUMMARY:
Background: Three-dimensional (3D) patient-specific anatomical model guidance is a reliable tool in obtaining accurate bony cuts, precise implant placement, and satisfactory surgical results. These can enhance surgeon's understanding of their patients' patho-anatomy also helping in precise preoperative planning. So, the hypothesis of this study is that, in the training of orthopaedic residency, 3D printed models reflecting the patient's individual process provide a a foresight and a perception of the bone pathologies and osseous relationships before orthopaedic intervention.

Methods: In this study, the investigators displayed our experience of creating realistic 3D models in orthopaedic surgical case scenarios to evaluate the perceptions of fellows in orthopaedic surgeon training. The investigators based our study on the comparision of the perception of residents who were presented with four-step carousel consisting of different scenarios as trauma (calcaneal fracture), deformity (hallux valgus), tumoral mass (sacral chondrosarcoma), and reconstructive procedure (multidisciplinary cancer surgery). The X-ray images, computed tomography (CT), and 1:1 solid models of the cases were included in each step. The orthopaedic residents were asked to compare their perception level of the actual scenarios in evaluating the effectiveness of each tool in terms of perceiving the orthopaedic problem, understanding the bone pathology, classification of diagnosis and preoperative data planning.

DETAILED DESCRIPTION:
2.1. Study Group The study group consisted of 11 orthopaedic residents of University Hospital. Ethics approval for this study was obtained from our university's Human Research Ethics Committee (18-5/41). The work has been reported in line with the STROCSS criteria.

2.2. Selection of the sample cases The patients were chosen from the MRI examinations of the ones who referred to same University Hospital Department of Orthopaedic and Traumatic Surgery for diagnosis and treatment between the year of 2016 and 2018. Selection criteria for the 4 cases was the involved patients (age: 18-62 years) who required orthopaedic surgery, had no previous orthopaedic nor traumatic operation, but on the other hand have bone pathology leading to deformity, fracture, and suitable radiological imaging results for modeling. 4 cases that could serve as an example for orthopaedic surgical procedures were determined with the consensus of experts in medical education, orthopaedic surgery and anatomy. The selected cases were turned into real scenarios with history, medical examination findings, and imaging methods. As data collection tool, descriptive grading scale was used to evaluate the perceptions of each of these imaging methods in terms of their usefulness in seeing the surgical problem, their efficiency in differential diagnosis and presurgical planning.

2.3.Image post-processing and segmentation Original CT images were converted into in Digital Imaging and Communications in Medicine (DICOM) format. Files were transferred to a separate workstation with Analyze 12.0 for post-processing and segmentation. Using free 3D Slicer (version 4.10.1) software, a smoothing filter was also applied to the segmented volume data to improve the surface quality of the model. The STL format for 3D printing was prepared.

2.4. Creating Life-size Patient-Specific 3D Model Mass Portal Pharaoh xd 20 printer was used due to its documented accuracy for producing high-resolution 3D models of orthopaedic cases from resin-based polymers.

2.5. Workshop Data collection shop A grading scale was developed for each case so that the residents were able to make a comparison.

1. The grading scale developed for the trauma case (calcaneus fracture) consisted of 16 items including the appearance, classification and planning of the fracture surgery.
2. The scale for the case of deformity (hallux valgus) contained 7 items of classification, questioning the degree of deformity and operation planning.
3. In the grading scale developed for the tumor case (chondrosarcoma), there were 13 items questioning the location, size, spread and neighboring pelvic structures.
4. In the scale for the reconstructive case (thorax localized tumor), there were 13 items questioning the location, size, spread and neighboring of intrathoracic structures, the occurrence of a postoperative defect, and the reconstructive method in the presence of a postoperative defect..

2.6. Survey A multi-item survey was prepared to assess fellow's perception of residency training. The survey utilized by our group, addressed the issues in understanding patient bone anatomy, seeing osseous pathology, independent decision-making, differential pathological diagnosis, plan on key surgical steps, and preparation for unexpected events. Residents who completed their examination in the stations evaluated each imaging method and answered the questions on a scale of 10. Scoring in the scale (1 - 10) describes 0 = very low and 10= the highest level.

2.7. Data collection Residents were asked to answer the grading scale by examining the X-ray, CT and the 3D model from the first station. In addition, opinions about the models were recorded and they were given an average of 10 minutes for each station.

2.8. Data Analysis Descriptive statistics and Friedman test were used for comparison analysis. Data were analyzed using IBM SPSS Statistics, version 24 (IBM Corp., Armonk, NY).

ELIGIBILITY:
Inclusion Criteria:Calcaneal fracture, Sacral tumors, Hallux valgus deformity, Mediastinal Tumors -

Exclusion Criteria:Tibial Fracture, Acetabular fracture, Femoral tumors, Pes planus

-

Ages: 24 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All assistants are men.
Study Population: The study group consisted of 11 orthopaedic residents of University Hospital.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Creating life-size patient-specific orthopaedic surgery cases model | The research took 12 months, 05.02.2020, Each participant spends 45 minutes for the survey.
  A multi-item survey was prepared to assess fellow's perception of residency training. The survey utilized by our group, addressed the issues in understanding patient bone anatomy, seeing osseous pathology, independent decision-making, differential pathological diagnosis, plan on key surgical steps, and preparation for unexpected events. Residents who completed their examination in the stations evaluated each imaging method and answered the questions on a scale of 10. Scoring in the scale (1 - 10) describes 0 = very low and 10= the highest level.Descriptive statistics and Friedman test were used for comparison analysis. Data were analyzed using IBM SPSS Statistics, version 24 (IBM Corp., Armonk, NY).

CONTACTS AND LOCATIONS:
Overall Officials: Yelda PINAR, Prof. Dr., Study Chair — Faculty of Medicine, Ege University
Locations (1):
- Ege University, Faculty of Medicine, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
In this study, we displayed our experience of creating realistic 3D models in orthopaedic surgical case scenarios to evaluate the perceptions of fellows in orthopaedic surgeon training. We based our study on the comparision of the perception of residents who were presented with four-step carousel consisting of different scenarios as trauma (calcaneal fracture), deformity (hallux valgus), tumoral mass (sacral chondrosarcoma), and reconstructive procedure (multidisciplinary cancer surgery). The X-ray images, computed tomography (CT), and 1:1 solid models of the cases were included in each step. The orthopaedic residents were asked to compare their perception level of the actual scenarios in evaluating the effectiveness of each tool in terms of perceiving the orthopaedic problem, understanding the bone pathology, classification of diagnosis and preoperative data planning.
Supporting Information: Study Protocol
Time Frame: Aim of this study, is also to show that the models can assist in the training of novice surgeons in complicated areas like trauma, deformity and cancer surgery. Yet another aim of the present study is to assess whether the 3D model could be more informative than standard X-ray and CT image visualizations in predicting the real outcome of the orthopaedic surgery cases.
Access Criteria: With the help of 3D printing technology, in this study, it is possible to implement and evaluate a well-structured real patient scenario setup for orthopaedic and traumatic surgery training. The orthopaedic intervention based on scenarios for residency is more original since there is no prior study including both model building and the evaluation of the perception created by the model. It can be used to improve the understanding of pathoanatomical changes of bone disease and to guide surgical strategy.